CLINICAL TRIAL: NCT06553690
Title: Impact of Brain Gym Therapy on Quality of Sleep Among Elderly People Attending Health Care Facilities
Brief Title: Brain Gym Therapy on Quality of Sleep Among Elderly People
Acronym: BG/E
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Shaban, dr, Cairo University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: braingym; HAP-13-S-001 (Other: Jouf university)
Record Dates: First submitted 2024-08-11; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Sleep Disorder; Insomnia; Cognitive Function Abnormal; Old Age; Debility; Brain Gym Therapy
Keywords: Brain Gym Therapy; Sleep Quality; Cognitive Exercise; Non-Pharmacological Intervention; Insomnia in Elderly
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders; Cognition Disorders; Frailty

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants receiving Brain Gym Therapy. (Experimental): Participants in this arm will undergo Brain Gym Therapy, which consists of a series of structured physical exercises designed to enhance cognitive function and promote relaxation.
  Interventions: Other: Brain Gym Therapy
- Participants receiving standard care without Brain Gym Therapy (No Intervention): standered care

INTERVENTIONS:
Other: Brain Gym Therapy — Brain Gym Therapy is a structured program of physical movements designed to enhance cognitive function, reduce stress, and promote relaxation. The therapy is based on the principle that specific physical activities can stimulate brain function and improve overall mental and physical well-being.
  Other Names: non
  Arms: Participants receiving Brain Gym Therapy.

SUMMARY:
This clinical trial aims to evaluate the impact of Brain Gym Therapy on the quality of sleep among elderly individuals attending healthcare facilities. The study will explore whether this non-pharmacological intervention can improve sleep quality, which is often compromised in the elderly population due to various health conditions and age-related changes. Participants will undergo Brain Gym Therapy sessions over a specified period, and their sleep quality will be assessed using validated sleep measurement tools. The findings may provide insights into alternative methods for enhancing sleep in older adults.

DETAILED DESCRIPTION:
This study investigates the effects of Brain Gym Therapy on the quality of sleep among elderly individuals who are receiving care at healthcare facilities. Brain Gym Therapy, a series of physical activities designed to enhance cognitive functions, has been hypothesized to positively influence sleep patterns by reducing stress, improving relaxation, and enhancing overall mental well-being.

The study will employ a randomized controlled trial design, with participants being randomly assigned to either an intervention group receiving Brain Gym Therapy or a control group receiving standard care without the therapy. The intervention will consist of structured Brain Gym exercises conducted by trained practitioners, focusing on movements that are believed to stimulate brain function and promote relaxation.

Participants will be elderly individuals aged 65 and above, attending healthcare facilities, and experiencing issues with sleep quality. Exclusion criteria will include individuals with severe cognitive impairments, those currently undergoing other sleep interventions, or those with contraindications to physical activity.

The primary outcome measure will be the quality of sleep, assessed using validated sleep questionnaires such as the Pittsburgh Sleep Quality Index (PSQI), alongside secondary outcomes including sleep latency, duration, and efficiency. Data will be collected at baseline, mid-intervention, and post-intervention, with follow-up assessments to determine the sustainability of any observed effects.

The study aims to contribute to the growing body of evidence supporting non-pharmacological interventions for sleep improvement in the elderly, potentially offering a viable alternative to medication for managing sleep disturbances in this population. Ethical approval has been obtained, and all participants will provide informed consent before participation

ELIGIBILITY:
Inclusion Criteria:

Elderly individuals aged 60 years and above. Attending healthcare facilities and able to participate in the study. Experiencing issues with sleep quality, as determined by a score of 5 or higher on the Pittsburgh Sleep Quality Index (PSQI).

Willing and able to provide informed consent. Physically capable of performing gentle physical exercises as part of Brain Gym Therapy

Exclusion Criteria:

Severe cognitive impairment or dementia that would impede understanding or participation in the intervention.

Current participation in another sleep intervention study. Presence of severe medical conditions that contraindicate physical activity (e.g., severe cardiovascular disease, musculoskeletal disorders).

Use of sleep medications that could confound the study results. Recent history (within the past 6 months) of major psychiatric disorders, including severe depression or anxiety.

Any condition that, in the opinion of the investigators, would make participation unsafe or not in the best interest of the participant.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2024-10-11 (Estimated); Study Completion 2024-10-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in Sleep Quality | Baseline, Week 4 (post-intervention), and Week 8 (follow-up)
  The primary outcome measure will assess the improvement in sleep quality among elderly participants who undergo Brain Gym Therapy compared to those receiving standard care. Sleep quality will be evaluated using the Pittsburgh Sleep Quality Index (PSQI), a validated and widely used instrument that measures various aspects of sleep including duration, latency, efficiency, disturbances, and subjective sleep quality. The PSQI score ranges from 0 to 21, with higher scores indicating poorer sleep quality.

REFERENCES:
- [Derived] Alanazi MA, Shaban M, Zaky ME. Impact of brain gym therapy on quality of sleep among older adults attending health care facilities. Geriatr Nurs. 2025 Jul-Aug;64:103431. doi: 10.1016/j.gerinurse.2025.103431. Epub 2025 Jun 27. PMID 40580820